CLINICAL TRIAL: NCT05398692
Title: Long COVID-19 Rehabilitation & Research Program
Brief Title: Long COVID-19 Rehabilitation & Recovery Research Program
Acronym: LC Rehab
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding exhausted.
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, William Stringer, md, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 032588-01
Record Dates: First submitted 2022-05-10; First posted 2022-06-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Post-Acute COVID-19 Syndrome; COVID-19
Keywords: Long COVID, COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Participants receive on site low to intermediate intensity exercise rehabilitation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- +/- PEM (Experimental): Patients with and without Post Exertional Malaise (PEM) will receive 10 weeks of on site low to moderate intensity exercise rehabilitation.
  Interventions: Other: On Site Exercise Rehabilitation

INTERVENTIONS:
Other: On Site Exercise Rehabilitation — The subject will receive on site standard pulmonary and exercise rehabilitation, educational instruction on balance and strength training, stretching, nutrition, hydration, pacing, proper breathing, small or mini-lectures, and information on relaxation techniques.

SUMMARY:
The purpose of the study is to assess the physiologic, immunologic, and mental health effects of an exercise and pulmonary rehabilitation program on patients with Long COVID-19 (LC).

DETAILED DESCRIPTION:
1.0 Objectives 1.1 Describe the purpose, specific aims, or objectives.

The purpose is to assess the physiologic, immunologic, and mental health effects of a rehabilitation program on patients with Long COVID-19 (LHC).

1.2 State the hypotheses to be tested.

Long COVID-19 Patients who enroll and complete a 10 week program of Physiologic and Psychological Rehabilitation will have reduced Long COVID-19 Symptoms, Improved Physical Status, Reduced Inflammatory Markers, and Augmented Psychological Well Being.

ELIGIBILITY:
Inclusion Criteria:

* Long COVID-19 Infection (Documented by PCR or patient report)
* Age >= 18 years old.
* At least 12 weeks since the initial COVID Infection.
* One or more of the following symptom/signs: Fatigue, Dyspnea, Exercise Intolerance, Post Exertional Malaise and/or Difficulty Breathing.
* Able to perform a cardiopulmonary exercise test.

Exclusion Criteria:

* Patients is not able to perform technically acceptable pulmonary function tests and symptom-limited cardiopulmonary cycle ergometry tests.
* Patients who desaturate to SpO2 <80% on screening incremental exercise testing.
* Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit or patients who are currently in a pulmonary rehabilitation program.
* Patients who have taken an investigational drug within one month or six half-lives (whichever is greater) prior to screening visit (Visit 1).
* Pregnant or nursing women.
* Women of childbearing potential who are not using a highly effective method of birth control. Female patients will be considered of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.
* Patients who are currently participating in another interventional study.
* Malignancy for which the patient has undergone resection, radiation therapy, or chemotherapy within the last 2 years
* Any other significant disease than COVID-19 which, in the opinion of the investigator, may i) put the patient at risk because of participation in the study, ii) influence the results of the study (e.g. Insulin or testosterone therapy, systemic corticosteroids, HIV, etc), iii) cause concern regarding the patient's ability to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in aerobic capacity (Peak Oxygen Uptake) at 10 weeks after rehabilitation comprehensive (normal intensity) pulmonary rehabilitation program. | 10 weeks
  Cardopulmonary - Exercise Outcomes.

SECONDARY OUTCOMES:
Short Form (SF-36) | 10 weeks
  Quality of Life - 36 Item Short Form Survey. 8 subdomains - Potential scores 0 to 100 (100 being best) in each domain.
Fatigue Severity Scale (FSS) | 10 weeks
  Change in a Fatigue Score - 9 questions -1 (strongly disagree) to 7 (strongly agree). Total score from 7 to 54. Lower numbers are better.
General Anxiety Disorder Screener (GAD-7) | 10 weeks
  Change in Anxiety scores - 7 questions. 0-Not at all to 3 Nearly Every Day - Scores from 0-21. Lower numbers are better.
Pittsburg Sleep Quality Score (PSQI) | 10 weeks
  Change in Sleep Quality Index - Scores from 0 to 42. Lower scores are better. A score > 5 indicates poor sleep quality.
Modified Medical Research Council Dyspnea Scale (mMRC) | 10 weeks
  Score ranges from 0 to 4. Lower scores are better.
Modified DePaul Assessment for Post-Exertional Malaise (DSQ-PEM) | 10 weeks
  Questions 6-10 Specific to PEM. All questions are Yes/No, No is best.
Patient Health Questionnaire (PHQ-9) | 10 weeks
  Change in Depression scores - 9 questions that are scored from 0-3. Total scores 0-27. Lower scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: William W Stringer, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbasi A, Gattoni C, Iacovino M, Ferguson C, Tosolini J, Singh A, Soe KK, Porszasz J, Lanks C, Rossiter HB, Casaburi R, Stringer WW. A Pilot Study on the Effects of Exercise Training on Cardiorespiratory Performance, Quality of Life, and Immunologic Variables in Long COVID. J Clin Med. 2024 Sep 20;13(18):5590. doi: 10.3390/jcm13185590. PMID 39337079
- [Derived] Abbasi A, Hansen N, Palade J, Paredes D, Meechoovet B, Van Keuren-Jensen K, Pirrotte P, Stringer WW. Serum extracellular vesicle RNA profiles in long COVID: insights from exercise-induced gene modulation. Sci Rep. 2026 Jan 26;16(1):3469. doi: 10.1038/s41598-025-23760-y. PMID 41588020